CLINICAL TRIAL: NCT04285437
Title: The Effects of Massage Therapy on Mental and Physical Development of Term Neonates and on Maternal Bonding.
Brief Title: The Effects of Massage Therapy on Term Neonates Development and on Maternal Bonding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Linh Dao Nguyen Phuong, Principal investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 414A/ĐHYD-HĐĐĐ
Record Dates: First submitted 2020-02-19; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Infant Development; Breastfeeding; Postnatal Depression
Keywords: infant massage
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- massage (Experimental): neonates are massaged by their mother during the first 2 months after birth.
  Interventions: Behavioral: infant massage
- control (No Intervention): neonates are not massaged.

INTERVENTIONS:
Behavioral: infant massage — Mother will be trained how to massage their babies by International Association of Infant Massage (IAIM) Certified Infant Massage Instructor, and then their babies will be massaged by themselves during the first 2 months after birth.
  Arms: massage

SUMMARY:
This study collects data from 2 groups of mother- term neonate pairs at the Neonatal Department of Children Hospital II, Ho Chi Minh City (in group M: neonates are massaged by their mothers during the first 2 months after birth, in group X: neonates are not massaged), and then, evaluates the effects of Massage Therapy on the mental and physical development of neonates and on maternal bonding (breast feeding, postnatal depression) during the first 2 months after birth.

DETAILED DESCRIPTION:
Infant Massage has been known for a long time, almost as far back as the first time it was recorded around 1800 BC. This was one of the original forms of medicine before the medical revolution broke out in the 1940s.

To date, more than 600 studies have been published on the effects of weight gain on massaged infants, primarily in preterm infants. In addition, the latest research also helps identify other effects such as shortening hospital time, better sleep, reducing pain, crying less, strengthen immunity, reducing bilirubin in neonates with jaundice.

On the other hand, the effect of the "parent direct massage for children" is also determined, the reports show an improvement in the parent-child interaction, increase breastfeeding, and reduce breastfeeding. The rate of postpartum depression reduced significantly.

Steps to proceed

* Step 1: Randomly select 2 groups of mother- term neonate pairs by letting every mother, who matching with eligibility criteria, draw 1 of 120 same color and size lotteries in which include 1 to 120 numbers randomly drawn from a web page https://stattrek.com/statistics/random-number-generator.aspx .

There are 2 groups of mother - term neonate pairs (60 pairs each):

* Group M: neonates are massaged by their mothers during the first 2 months after birth. Mothers in this group will be given instructions on breastfeeding, and massage therapy (by principal investigator as International Association of Infant Massage Certified Instructor) in 2 days before discharge, and mothers will record "Parenting Dairy" form (The diary includes the number of defecation times, the number of spitting up times, the number of crying times over 15 minutes, the number of massage times, and the sleep time during the day)
* Group X: neonates are not massaged. Mothers in this group will be given instructions on breastfeeding only, and they will record "Dairy of taking care baby" form like the other group.

  * Step 2: At 1 day after discharge, the investigator make a phone call with mothers of group M to track and remind them massage for their babies.
  * Step 3: At the time of 10 days before the baby turn 1 month - old and 2 month - old, the investigator make a phone call with mothers in both groups to track and remind massage for children (group M), as well as the record "Parenting Dairy" (both groups)
  * Step 4: At the time the child turn 1 month - old and 2 month - old, the investigator make a home visit to both groups, let mothers perform Edinburgh Postnatal Depression Scale, collect data from "Parenting Dairy", assess the height - weight - head circle of the babies.

ELIGIBILITY:
Inclusion Criteria: Group of mother and neonate at Neonatal Department of Children Hospital II, Ho Chi Minh City

* neonate: full term, not low birth weight, 0 - 15 days of age, diagnosed with one of the following conditions and has been treated stably: uncomplicated neonatal infection, uncomplicated pneumonia, non umbilical cord infection, uncomplicated neonatal jaundice
* mother: live in Ho Chi Minh City

Exclusion Criteria: If the mother or neonate has the criteria to eliminate:

* Mother with mental illness, developmental disorder, prenatal depression, not directly caring for children.
* Neonate with multiple deformities, asphyxia, severe jaundice with complication, cow's milk allergy, heart/ lung/central nervous system defects.

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
The rate of pairs that have Edinburgh Postnatal Depression Scale scored > 12 | at the day baby turns 1 month of age
  When home visiting, the investigator let the mother do Edinburgh Postnatal Depression Scale
The rate of pairs that have Edinburgh Postnatal Depression Scale scored > 12 | at the day baby turns 2 month of age
  When home visiting, the investigator let the mother do Edinburgh Postnatal Depression Scale
Change of the number of crying times over 15 minutes at 2 month - old - infant | 2 months after birth
  When home visiting, the investigator collect from "Parenting Dairy"
The rate of pairs that have breastfeeding | at the day baby turns 1 month of age
  When home visiting, the investigator collect from "Parenting Dairy"
The rate of pairs that have breastfeeding | at the day baby turns 2 month of age
  When home visiting, the investigator collect from "Parenting Dairy"

SECONDARY OUTCOMES:
The mean of Edinburgh Postnatal Depression Scale | at the day baby turns 1 month of age
  When home visiting, the investigator let the mother do Edinburgh Postnatal Depression Scale
The mean of Edinburgh Postnatal Depression Scale | at the day baby turns 2 month of age
  When home visiting, the investigator let the mother do Edinburgh Postnatal Depression Scale
Change of the number of defecation times at 2 month - old - infant | 2 months after birth
  When home visiting, the investigator collect from "Parenting Dairy"
Change of the number of spitting up at 2 month - old - infant | 2 months after birth
  When home visiting, the investigator collect from "Parenting Dairy"
Change of weight at 2 month - old - infant | 2 months after birth
  When home visiting, the investigator assess the weight of infant
Change of height at 2 month - old - infant | 2 months after birth
  When home visiting, the investigator assess the height of infant
Change of head circle at 2 month - old - infant | 2 months after birth
  When home visiting, the investigator assess the head circle of infant

CONTACTS AND LOCATIONS:
Overall Officials: Tuan Le Minh, Ph.D, MD, Study Chair — Research Department, UMP
Locations (1):
- University of Medicine and Pharmacy, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No